CLINICAL TRIAL: NCT01544127
Title: Motivational Interviewing to Prevent Suicide in High Risk Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-20-11S; IK2CX00064 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Suicidal Ideation; Treatment Engagement
Keywords: Veterans; Motivational Interviewing; Inpatients; Suicide, Attempted
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MI-SI+TAU (Experimental): Motivational Interviewing to Address Suicidal Ideation
  Interventions: Behavioral: MI-SI+TAU
- MI-SI-R+TAU (Experimental): Motivational Interviewing to Address Suicidal Ideation Revised
  Interventions: Behavioral: MI-SI-R+TAU
- TAU Alone (Other): Treatment as usual
  Interventions: Other: TAU Alone

INTERVENTIONS:
Behavioral: MI-SI+TAU — MI-SI focuses on exploring and resolving ambivalence about living. It consists of 1 or 2 in-person MI-SI sessions (50 mins.) on an inpatient unit, plus a telephone follow-up MI-SI session (30-50 mins)
  Other Names: Motivational Interviewing to Address Suicidal Ideation
  Arms: MI-SI+TAU
Behavioral: MI-SI-R+TAU — MI-SI-R focuses on resolving ambivalence about living. It consists of 1 or 2 in-person MI-SI sessions (50 mins.) on an inpatient unit, plus a telephone follow-up MI-SI session (30-50 mins)
  Other Names: MI-SI Revised
  Arms: MI-SI-R+TAU
Other: TAU Alone — Inpatient treatment includes medication management, case management, meals and a bed, milieu therapy consisting of creative and social activities, and a safety plan. Some families of veterans also received education to create a supportive home environment. As part of Veterans Health Administration (VHA) suicide prevention policy, the care of suicidal patients is also overseen by a local Suicide Prevention Coordinator and case managers.
  Other Names: Treatment as usual
  Arms: TAU Alone

SUMMARY:
The purpose of study is to test the efficacy of an adaptation of Motivational Interviewing to Address Suicidal Ideation (MI-SI) on the severity of suicidal ideation in psychiatrically hospitalized Veterans at high risk for suicide.

DETAILED DESCRIPTION:
Veterans who receive health care from the VA are at elevated risk for suicide, and the number of Veterans at high risk may be growing. Although the months following discharge from psychiatric hospitalization are a period of acute risk for Veterans, there is a dearth of empirically supported treatments tailored to psychiatric inpatients and no studies examining treatments for psychiatrically hospitalized Veterans. This randomized controlled trial will test the efficacy of an adaptation of Motivational Interviewing to Address Suicidal Ideation (MI-SI) on the severity of suicidal ideation in psychiatrically hospitalized Veterans at high risk for suicide. Participants will be recruited from the Acute Psychiatric Inpatient Unit at the Syracuse VA Medical Center. To meet high-risk criteria, Veterans must score over two on the Scale for Suicidal Ideation (SSI), which is prospectively predictive of death by suicide. Participants will complete a screening assessment to confirm eligibility and a baseline assessment of risk factors for suicide. They will be randomized to receive Motivational Interviewing to Address Suicidal Ideation (MI-SI) or a revised version (MI-SI-R) plus treatment as usual (TAU), or TAU alone. The MI-SI groups will receive two sessions of MI-SI during hospitalization and one telephone booster session after discharge. Participants in all conditions will be asked to complete telephone follow-up interviews at 1, 3, and 6 months after discharge. Change in the severity of suicidal ideation will be measured using the SSI.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status,
* admitted to psychiatric inpatient unit,
* age 18 and over,
* English speaking,
* able to understand the study and provide informed consent,
* clinically cleared to participate by unit staff,
* receive health care from a VHA facility in upstate New York
* at increased risk for suicide (Scale for Suicidal Ideation [SSI] > 2)

Exclusion Criteria:

* current psychosis,
* current mania,
* dementia,
* prisoner status,
* being inaccessible
* being discharged from the unit less than 48 hours after being identified by study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-07-30 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Britton, PhD MS, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Britton PC, Conner KR, Chapman BP, Maisto SA. Motivational Interviewing to Address Suicidal Ideation: A Randomized Controlled Trial in Veterans. Suicide Life Threat Behav. 2020 Feb;50(1):233-248. doi: 10.1111/sltb.12581. Epub 2019 Aug 8. PMID 31393029

RESULTS

PARTICIPANT FLOW:
Groups:
- MI-SI: Motivational interviewing to address suicidal ideation (MI-SI) is an adaptation of motivational interviewing that is focused on exploring and resolving ambivalence about living.
- MI-SI-R: Motivational interviewing to address suicidal ideation revised (MI-SI-R) is an adaptation of motivational interviewing that is focused on resolving ambivalence about living.
- VA TAU: Treatment as usual is standard treatment received during acute psychiatric hospitalization in a Department of Veterans Affairs (VA) medical center and after discharge.
Period: Overall Study
Arm/Group | MI-SI | MI-SI-R | VA TAU
Started | 33 | 33 | 66
Completed | 22 | 27 | 52
Not Completed | 11 | 6 | 14
Not completed — Lost to Follow-up | 4 | 2 | 9
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Discharged out of catchment area | 1 | 1 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Jail or Prison | 1 | 1 | 2
Not completed — Became Psychotic | 1 | 0 | 0
Not completed — Researcher withdrew | 1 | 0 | 0
Not completed — Went active duty | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- MI-SI+TAU: Motivational Interviewing to Address Suicidal Ideation (MI-SI)
  MI-SI focuses on exploring and resolving ambivalence about living. It consist of 1 or 2 in-person MI-SI sessions (50 mins.) on an inpatient unit, plus a telephone follow-up session (30-50 mins)
- MI-SI-R+TAU: Motivational Interviewing to Address Suicidal Ideation Revised (MI-SI-R)
  MI-SI-R focuses on resolving ambivalence about living. It consists of 1 or 2 in-person MI-SI sessions (50 mins.) on an inpatient unit, plus a telephone follow-up MI-SI session (30-50 mins)
- Treatment as Usual (TAU): Treatment as Usual (TAU)
  TAU consisted of standard inpatient treatment that includes medication management, case management, meals and a bed, and milieu therapy consisting of creative and social activities. Some families of veterans also received education to create a supportive home environment. Suicidal patients also completed a safety plan prior to discharge, and their care was overseen by a local Suicide Prevention Coordinator and case managers.
- Total: Total of all reporting groups
Arm/Group | MI-SI+TAU | MI-SI-R+TAU | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 33 | 33 | 66 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.61 (12.69) | 43.91 (12.44) | 46.03 (12.77) | 45.64 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 8 | 14
  Male | 30 | 30 | 58 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 32 | 33 | 64 | 129
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 5 | 5 | 8 | 18
  White | 25 | 25 | 52 | 102
  More than one race | 0 | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Marital Status [Count of Participants; unit: Participants]
  Married | 13 | 9 | 22 | 44
  Divorced/Separated | 9 | 15 | 33 | 57
  Never Married | 8 | 7 | 10 | 25
  Widowed | 3 | 2 | 1 | 6
Employment [Count of Participants; unit: Participants]
  Part/Fulltime/Self-Employed | 4 | 6 | 14 | 24
  Student/Homemaker | 0 | 0 | 2 | 2
  Unemployed | 11 | 6 | 18 | 35
  Disabled/Retired | 18 | 21 | 31 | 70
  Other | 0 | 0 | 1 | 1
Years of Service [Mean (Standard Deviation); unit: years] | 6.21 (7.05) | 5.82 (4.82) | 7.09 (6.78) | 6.55 (6.40)
Era [Count of Participants; unit: Participants]
  Post 9/11 (2001-Present) | 7 | 13 | 17 | 37
  Desert Storm/Shield (1990-2001) | 2 | 3 | 5 | 10
  Post-Vietnam Peace (1975-1990) | 9 | 6 | 16 | 31
  Vietnam War (1964-1975) | 6 | 1 | 5 | 12
  Post-Korea Peace (1955-1964) | 0 | 0 | 2 | 2
  Multiple Eras | 9 | 10 | 21 | 40
Deployed to Combat Zone [Count of Participants; unit: Participants] | 15 | 17 | 30 | 62
Scale for Suicidal Ideation (SSI) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 38, with higher scores indicating more severe suicidal ideation.
  units on a scale
    Current (week before hospitalization) | 23.27 (8.33) | 20.06 (7.73) | 20.54 (8.64) | 21.11 (24.85)
    Worst Point | 26.75 (8.50) | 25.76 (8.81) | 23.45 (9.07) | 24.85 (8.92)
Columbia- Suicide Severity Rating Scale (C-SSRS): Suicide Attempt Last Month [Count of Participants; unit: Participants] | 6 | 7 | 17 | 30
C-SSRS: Lifetime Suicide Attempts [Mean (Standard Deviation); unit: events] | 2.85 (3.44) | 1.84 (2.81) | 1.24 (1.66) | 1.80 (2.57)
Ohio State University Traumatic Brain Injury Identification Method (TBI-ID): Loss of Consciousness [Mean (Standard Deviation); unit: events]
  #Times | 2.03 (2.23) | 1.91 (2.11) | 1.18 (1.71) | 1.58 (1.98)
  # Times >= 30 mins | 0.42 (0.66) | 0.21 (0.42) | 0.17 (0.41) | 0.24 (0.50)
TBI-ID: Loss of Consciousness Before 15 Years of Age [Count of Participants; unit: Participants] | 11 | 12 | 12 | 35
TBI-ID: Worst TBI [Mean (Standard Deviation); unit: units on a scale] — Scores range from 1 to 5, with higher scores indicating more severe TBI.
  units on a scale | 3.00 (1.06) | 2.70 (1.10) | 2.44 (1.18) | 2.64 (1.15)
Patient Health Questionnaire (PHQ-9): Depression [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
  units on a scale | 18.54 (4.29) | 18.12 (4.74) | 17.92 (5.28) | 18.13 (4.88)
Posttraumatic Stress Disorder (PTSD) Checklist Civilian Version (PCL-C) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 17 to 85, with higher scores indicating more severe PTSD symptoms.
  units on a scale | 60.12 (11.07) | 58.39 (12.73) | 56.89 (13.35) | 58.08 (12.64)
Beck Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 63, with higher score indicating more severe anxiety symptoms.
  units on a scale | 26.09 (10.72) | 27.21 (12.72) | 28.24 (10.20) | 26.91 (11.08)
Alcohol Use Disorders Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 40, with higher scores indicating hazardous alcohol use.
  units on a scale | 14.54 (11.50) | 9.67 (10.19) | 14.48 (12.53) | 12.80 (11.81)
Drug Abuse Screening Test (DAST) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 10, with higher score indicating more hazardous non-alcohol drug use.
  units on a scale | 2.58 (2.90) | 2.85 (3.38) | 3.02 (3.31) | 2.86 (3.21)
Addiction Severity Index (ASI) (past 28 days) [Mean (Standard Deviation); unit: days]
  Any Mental Health Inpatient Days | 0.27 (1.15) | 2.82 (7.38) | 2.39 (6.32) | 1.97 (5.87)
  Any Mental Health Outpatient Days | 2.58 (4.47) | 2.83 (4.43) | 3.58 (5.50) | 2.82 (4.43)
  Psychiatric Medication | 14.82 (12.87) | 18.70 (12.61) | 17.20 (12.82) | 16.98 (12.76)
  Medical Medication | 16.15 (12.96) | 14.00 (14.00) | 14.45 (13.36) | 14.77 (13.35)
  Substance Abuse Medication | 1.85 (6.09) | 0.03 (0.17) | 2.14 (7.08) | 1.54 (5.89)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suicidal Ideation
Description: The number of participants with suicidal ideation and severity of suicidal ideation was measured using the Scale for Suicidal Ideation (SSI) at 1, 3, and 6 months after discharge. Scores range from 0-38, with scores of 1 or greater indicating the presence of suicidal ideation.
Time Frame: 6 months
Population: Analytical sample consists of participants who completed at least one follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- TAU Alone: Treatment as usual
  TAU: Inpatient treatment includes medication management, case management, meals and a bed, milieu therapy consisting of creative and social activities, and a safety plan. Some families of veterans also received education to create a supportive home environment. As part of Veterans Health Administration(VHA) suicide prevention policy, the care of suicidal patients is also overseen by a local Suicide Prevention Coordinator and case managers.
Arm/Group | MI-SI+TAU | MI-SI-R+TAU | TAU Alone
Number analyzed (Participants) | 28 | 31 | 63
Participants
  1 Month: number analyzed (Participants) | 24 | 27 | 56
  1 Month | 16 | 19 | 38
  3 Months: number analyzed (Participants) | 23 | 26 | 55
  3 Months | 17 | 16 | 42
  6 Months: number analyzed (Participants) | 21 | 28 | 52
  6 Months | 13 | 18 | 40
Statistical Analysis 1: Comparison: MI-SI+TAU vs MI-SI-R+TAU vs TAU Alone; MI-SI + TAU and MI-SI-R + TAU vs. TAU Alone A hurdle model was used to examine the effect of the experimental interventions on the presence of suicidal ideation and the severity of suicidal ideation among those with it. These analyses examined the presence of suicidal ideation in the combined MI-SI + TAU and MI-SI-R + TAU treatment group; Test type: Superiority; p = .054, Zero-Inflated Poisson — A priori, analyses were proposed to be one-sided, with p set at 0.05; Analysis adjusted for severity of worst TBI experience and used a robust standard error that was clustered on participants; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.31 to 1.12], Standard Error of Mean 0.19 — OR was calculated for number of participants with suicidal ideation. Analyses were one-sided, but two-sided confidence intervals for the OR are reported
Statistical Analysis 2: Comparison: MI-SI+TAU vs TAU Alone; MI-SI+TAU vs. TAU Alone; Test type: Superiority; p = 0.12, Zero-Inflated Poisson — A priori, analyses were proposed as one-sided, with p set at 0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.26 to 1.40], Standard Error of Mean 0.26 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: MI-SI-R+TAU vs TAU Alone; MI-SI-R + TAU vs. TAU Alone; Test type: Superiority; p = 0.08, Zero-Inflated Poisson — A priori, analyses were proposed as one-sided, with p set at 0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.28 to 1.24], Standard Error of Mean 0.22 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Severity of Suicidal Ideation Among Those With It
Description: Severity of suicidal ideation was measured by the Scale for Suicidal Ideation at 1, 3, and 6 months after discharge. Scores range from 0 to 38, with higher scores indicating more severe suicidal ideation.
Time Frame: 6 months
Population: Analyses were limited to the participants who reported suicidal ideation over follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MI-SI+TAU | MI-SI-R+TAU | TAU Alone
Number analyzed (Participants) | 25 | 27 | 54
score on a scale
  1 month: number analyzed (Participants) | 16 | 19 | 38
  1 month | 16.94 (9.05) | 14.26 (9.70) | 14.21 (9.62)
  3 months: number analyzed (Participants) | 17 | 16 | 40
  3 months | 8.88 (9.05) | 15.25 (9.39) | 12.74 (8.57)
  6 months: number analyzed (Participants) | 13 | 18 | 40
  6 months | 18.15 (10.52) | 16.89 (9.18) | 15.45 (10.06)
Statistical Analysis 1: Comparison: MI-SI+TAU vs MI-SI-R+TAU vs TAU Alone; MI-SI + TAU vs. MI-SI-R + TAU vs. TAU Alone A hurdle model was used to examine the effect of the experimental interventions on the presence/absence of suicidal ideation and the severity of suicidal ideation among those with it. These analyses examined the severity of suicidal ideation among participants with suicidal ideation in the combined MI-SI + TAU and MI-SI-R + TAU treatment group; Test type: Superiority; p = 0.30, Zero-Inflated Poisson — A priori, analyses were proposed to be one-sided, with p set at 0.05; A robust standard error clustered on participants was used; Beta = 0.06, Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: MI-SI+TAU vs TAU Alone; MI-SI vs. TAU Alone; Test type: Superiority; p = 0.23, Zero-Inflated Poisson — A priori, analyses were proposed to be one-sided, with p set at 0.05; A robust standard error clustered on participants was used; Beta = 0.09, Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: MI-SI-R+TAU vs TAU Alone; MI-SI-R vs. TAU Alone; Test type: Superiority; p = 0.46, Zero-Inflated Poisson — A priori, analyses were proposed to be one-sided, with p set at 0.05; A robust standard error clustered on participants was used; Beta = 0.01, Standard Error of Mean 0.13

3. Secondary Outcome: Number of Participants With Two Outpatient Mental Health or Substance Treatment Sessions
Description: Treatment engagement was measured using the Treatment Services Review-6 (TSR-6) at 1 month after discharge.
Time Frame: 1 month
Population: Analyses were limited to participants who were immediately discharged to outpatient treatment.
Measure: Count of Participants; unit: Participants
Groups:
- TAU Alone: Treatment as usual
  TAU: Inpatient treatment includes medication management, case management, meals and a bed, milieu therapy consisting of creative and social activities, and a safety plan. Some families of veterans also received education to create a supportive home environment. As part of VHA suicide prevention policy, the care of suicidal patients is also overseen by a local Suicide Prevention Coordinator and case managers.
Arm/Group | MI-SI+TAU | MI-SI-R+TAU | TAU Alone
Number analyzed (Participants) | 21 | 25 | 41
Participants | 16 | 17 | 31
Statistical Analysis 1: Comparison: MI-SI+TAU vs TAU Alone; MI-SI + TAU vs. TAU Alone; Test type: Superiority; p = 0.96, Regression, Logistic — A priori, p was set at 0.01 for multiple comparisons; Odds Ratio (OR) = 1.03, 0.95% CI 2-sided [0.30 to 3.54], Standard Error of Mean 0.65
Statistical Analysis 2: Comparison: MI-SI-R+TAU vs TAU Alone; MI-SI-R + TAU vs. TAU Alone; Test type: Superiority; p = 0.50, Regression, Logistic — A priori, p was set at 0.01 for multiple comparisons; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.23 to 2.06], Standard Error of Mean 0.38

4. Other Pre Specified Outcome: Number of Participants With a Suicide Attempt
Description: Presence of a suicide attempt was measured with the Columbia Suicide Severity Rating Scale (C-SSRS) at 1, 3, and 6 months after discharge.
Time Frame: 1, 3, and 6 months
Population: All participants were entered into analyses and censored at suicide attempt or the last follow-up assessment. Follow-up assessments were completed by 122 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | MI-SI+TAU | MI-SI-R+TAU | TAU Alone
Number analyzed (Participants) | 28 | 31 | 63
Participants
  1 Month | 2 | 1 | 5
  3 Months: number analyzed (Participants) | 25 | 28 | 54
  3 Months | 2 | 1 | 1
  6 Months: number analyzed (Participants) | 20 | 26 | 47
  6 Months | 2 | 0 | 2
Statistical Analysis 1: Comparison: MI-SI+TAU vs TAU Alone; MI-SI + TAU vs. TAU Alone; Test type: Superiority; p = 0.31, Log Rank — A priori, p was set at 0.01 for multiple comparisons; Cox Proportional Hazard = 1.69, 95% CI 2-sided [0.59 to 4.88], Standard Error of Mean 0.91
Statistical Analysis 2: Comparison: MI-SI-R+TAU vs TAU Alone; MI-SI-R vs. TAU Alone; Test type: Superiority; p = 0.24, Log Rank — A priori, p was set at 0.01 for multiple comparisons; Cox Proportional Hazard = 0.49, 95% CI 2-sided [0.10 to 2.31], Standard Error of Mean 0.39
Statistical Analysis 3: Comparison: MI-SI+TAU vs MI-SI-R+TAU; MI-SI-R + TAU vs. MI-SI + TAU Because the impact of MI-SI + TAU and MI-SI-R + TAU were in different directions when compared to TAU Alone, they were compared. For this analysis, the null hypothesis was that the revisions did not change the impact of MI-SI + TAU; Test type: Superiority; p = 0.10, Log Rank — A priori, p was set at 0.01 for multiple comparisons; Cox Proportional Hazard = 0.29, 95% CI 2-sided [0.06 to 1.43], Standard Error of Mean 0.23

ADVERSE EVENTS:
Time Frame: 6 months
Description: For this study, serious adverse events were death and other life-threatening events including suicide attempts and accidental overdose. Adverse events were suicidal ideation or psychiatric symptoms that led to an Emergency Department visit and/or hospitalization.
Arm/Group | MI-SI+TAU | MI-SI-R+TAU | TAU Alone
All-Cause Mortality (participants affected / at risk) | 1/33 | 0/33 | 0/66
Serious Adverse Events (participants affected / at risk) | 7/33 | 3/33 | 12/66
Other Adverse Events (participants affected / at risk) | 10/33 | 10/33 | 21/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MI-SI+TAU (N=33) | MI-SI-R+TAU (N=33) | TAU Alone (N=66)
Suicide Attempt (Psychiatric disorders) | 5 (6) | 3 (4) | 10 (11)
Accidental Overdose (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Death (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MI-SI+TAU (N=33) | MI-SI-R+TAU (N=33) | TAU Alone (N=66)
Suicidal ideation (Psychiatric disorders) | 9 (11) | 8 (10) | 19 (24) — that led to Emergency Department visit and/or hospitalization.
Psychiatric Symptoms (Psychiatric disorders) | 2 (2) | 3 (4) | 5 (5) — that led to Emergency Department visit and/or hospitalization

LIMITATIONS AND CAVEATS:
Due to theoretical and empirically supported changes to motivational interviewing that were published during the trial, we changed the intervention mid-trial leading to small numbers of participants in the experimental conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT01544127/Prot_SAP_000.pdf